CLINICAL TRIAL: NCT04895579
Title: Boosting Immune Response With Copanlisib in Locally Advanced Unresectable Non-Small Cell Lung Cancer Receiving Durvalumab, A Phase Ib Study
Brief Title: Lung Cancer With Copanlisib and Durvalumab
Acronym: LCD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhonglin Hao (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Zhonglin Hao, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-LUN-119-PMC
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Stage 3A, 3B; Chemoradiation therapy; Durvalumab consolidation/maintenance; Copanlisib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; copanlisib

STUDY DESIGN:
Intervention Model Description: Dose finding cohort and dose expansion cohort up to 18 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib (30-60mg iv) (Experimental): Patients in the group will receive Durvalumab at 10mg/kg (IV infusion on days 1 and 15, q28 days or 1500mg day 1 q28d). They will also receive Copanlisib ranging from 30mg to 60mg (IV infusion on days 1 and 15, q 28 days).
  Interventions: Drug: Durvalumab; Drug: Copanlisib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be delivered at 10mg/kg via IV infusion at days 1 and 15 every 28 days or 1500 mg on D1, q4w.
  Other Names: Imfinzi
Drug: Copanlisib — Copanlisib will be delivered at various doses (30-60mg/kg) via IV infusion at days 1 and 15 every 28 days.
  Other Names: Aliqopa

SUMMARY:
The current study focuses on unresectable stage III non-small cell lung cancer (NSCLC) patients who are starting Durvalumab consolidation after concurrent chemoradiation with a goal of cure. The overall hypothesis of this study is that the addition of Copanlisib to Durvalumab will be well-tolerated at a biweekly schedule. It will test whether the addition of Copanlisib to Durvalumab can overcome resistance to Durvalumab.

DETAILED DESCRIPTION:
Treatment will be administered in outpatient settings. Durvalumab will be administered as infusion intravenously once every two weeks on D1 and D15, every 28 days (10 mg/Kg based on body weight) or 1500mg on D1 every 28 days. Copanlisib will be given as infusion intravenously on D1, D15 in a 28-day cycle (flat dose). The starting dose of Copalisib will be 60 mg D1 and D15. It will be reduced to 45 mg for the first dose reduction and to 30 mg for the second dose reduction. The Durvalumab dose will remain constant when Copanlisib is reduced.

Once the appropriate dose is determined, e.g. Copanlisib 60 mg iv d1, 15, q4w, in the dose-finding phase, this will become the recommended dose for the dose-expansion phase. Patients will be treated at the dose-expansion phase to increase our understanding of pharmacokinetics and to confirm safety as well as initial efficacy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (e.g., adenocarcinoma, squamous cell) deemed unresectable or inoperable who have received concurrent chemoradiation.
* Durvalumab will be started as consolidation therapy
* Have at least one measurable lesion.
* ECOG performance status ≤2.
* Adequate organ and marrow function.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Mixed Non-small cell and small cell histology; known EGFR and/or ALK driver mutations.
* Treated with sequential chemoradiation therapy.
* Autoimmune disease, such as rheumatoid arthritis, systemic lupus erythematosus, requiring systemic treatment with immunosuppressant in the past two years.
* Patients who are receiving any other investigational agents orally or intravenously.
* Systemic steroid for other purpose exceeding 10 mg prednisone a day except local injection at the discretion of the investigator.
* Solid organ or bone marrow transplant recipients.
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function.
* Patients with uncontrolled inter-current illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements and patients with seizure disorder not well controlled.
* Received live vaccine in the past 4 weeks.
* Pregnant or breast-feeding/lactating women.
* Receiving medications prohibited by the study.
* New York Heart Association Class 3 or above.
* Myocardial infarction within the last 6 months.
* Unstable angina.
* Venous thromboembolism within last 3 months.
* Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks.
* Proteinuria of ≥ CTCAE Grade 3 or estimated by urine protein: creatinine ratio > 3.5
* Major surgeries within the last 28 days.
* Any illness or medical conditions that are unstable or could jeopardize the safety of patients and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
  The number of dose limiting toxicities will be counted for each cohort.

SECONDARY OUTCOMES:
Objective Response Rate | approximately 10 years
  The objective response rate is evaluated by iRECIST 1.1, which includes all patients with partial response (iPR) or complete response (iCR).
Progression-Free Survival | approximately 10 years
  Progression-free survival (PFS) is defined as the time interval between the date patients are started on Copanlisib treatment to the date of disease progression, death or last follow-up, whichever occurs first. Patients who are intolerant to treatment and removed from study by the principal investigator or withdraw from the study will be treated as censored data for the PFS analysis.
Duration of Response | approximately 10 years
  Duration of response (DOR) is defined as the time interval between the initial response to therapy and subsequent disease progression or relapse. Non-responders will be assigned a DOR equal to zero.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonglin Hao, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No